CLINICAL TRIAL: NCT02917382
Title: Evolution of Nutritional Status, Metabolic, Functional and Clinical Outcomes in Patients Undergoing Liver Transplantation
Brief Title: Evolution and Clinical Outcomes in Patients Undergoing Liver Transplantation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Maria Isabel Toulson Davisson Correia, PHD, Federal University of Minas Gerais
Other Study IDs: FU Minas Gerais
Record Dates: First submitted 2016-08-11; First posted 2016-09-28 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Liver Disease; Nutrition Disorders
MeSH Terms: conditions — Liver Diseases; Nutrition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Waiting list for liver transplant: Patients on the waiting list for liver transplant treated at ambulatory liver transplant of Hospital of Clinics of the Federal University of Minas Gerais
- Undergoing liver transplantation: Patients undergoing liver transplantation treated at ambulatory liver transplant of Hospital of Clinics of the Federal University of Minas Gerais

SUMMARY:
Liver transplantation (LTx) is the standard treatment used in the final stage of chronic or acute liver failure. The success for the LT depends on many factors. One of the factors related to morbidity and mortality of these patients is malnutrition. Patients on the waiting list for LTx are increased risk of malnutrition and metabolic disorders that may be associated with decreased functional capacity, change in resting energy expenditure cardiac autonomic dysfunction. These conditions may influence the results both before and after transplantation, as the clinical outcome and complications present in the postoperative period. Therefore, this study aims to characterize and relate nutritional status, metabolic, functional and clinical outcomes in the recent postoperative patients undergoing liver transplantation. It is an observational, prospective study based on four evaluations: the first will be conducted while the patient is awaiting transplantation; and after insertion of the graft, patients will be evaluated between the 1nd and 3th postoperative day, between 5 and 7 days and at discharge from hospital.

In the late post-transplant, there is the action of immunosuppressive drugs, largely responsible for increased survival, but also on the other hand, are responsible for important nutritional and metabolic disorders. Metabolic complications such as hyperkalemia, hypertension, diabetes mellitus and overweight have been described. Thus, due to the high incidence of these complications, alternative options, such as lowering the dose of immunosuppressive drugs, have been fully explored, particularly as regards association with the viability of the graft. However, few studies have evaluated whether there is change in the incidence of metabolic disorders, cited above, in relation to the different doses of immunosuppressive drugs. Furthermore these metabolic complications will be evaluated in the late post-transplant period.

DETAILED DESCRIPTION:
This study was carried out at the Alfa Institute of Gastroenterology, Hospital of Clinics, Universidade Federal of Minas Gerais (UFMG). The research protocol was approved by the UFMG Ethics Committee. Patients with indication for liver transplantation, aged over 20 years who regularly attended the Liver Outpatient Transplant Clinic were included after having agreed and signed the informed consent form. Patients on the waiting list for a double or re-transplant were excluding conditions.

Nutritional status was provided by the Subjective Global Assessment (SGA), adapted for patients on the waiting list for liver transplantation is based on clinical history and physical examination, as well as the presence of existing conditions such as encephalopathy, chronic or recurrent infection, varicose veins and renal function.

Anthropometric evaluation was comprised of weight, height, body mass index (BMI), triceps and subscapular skinfold thickness (TSF and SSF respectively, measured with the Lange Skinfold Caliper - Cambridge Scientific Industries Inc., Cambridge, MD, USA), and arm muscle area (AMA). To minimize practical variability, the average of three consecutive measurements was recorded.

Functional parameters were evaluated by Handgrip strength (HS), 6-minute walk test (6MWT) and heart frequency variability (HFV). HS was assessed with the Jamar Handgrip Dynamometer (Preston, Jackson, MI, USA) using the non-dominant arm, and the mean of three measurements was determined. The 6MWT was performed indoors, in a 30m long, flat corridor with an adequate surface and the gait speed during the 6MWT was collected. The HRV was assessed using short-term evaluation. The heart rate recording was acquired by RS800 CX (Polar, Finland) and a 5-min stable cardiac recording was analyzed to assess the time domain (SD of all normal-to-normal interval [SDNN]).

Bioelectrical impedance analysis (Quantum X - RJL Systems, Inc., Clinton Township, Michigan) was used to determine body composition. Measurements were made with patients lying in bed with 4 electrodes attached to the dorsum of the right hand and foot. Phase angle (PA), fat mass (FM - kg), fat free mass (FFM, kg), total body water (TBW - L), intracellular water (ICW - L) and extracellular water (ECW - L), were evaluated.

Resting Energy Expenditure - REE was measured by indirect calorimetry using Quark RMR® (Cosmed, Rome, Italy). The energy balance (EB) was obtained by subtracting the total energy expenditure from the total caloric intake (TCI). The total energy expenditure (TEE) was obtained by multiplying the 24-hour REE by the calculated activity factor (AF), which was based on the description of the patients' daily activities and the corresponding computed values of metabolic equivalents (METs). Food intake was assessed by a 3-day food record (Avanutri Online® (Avanutri Equipamentos de Avaliação Ltda, Rio de Janeiro, Brazil).

Clinical and other variables - Age, sex, etiology, severity of liver disease by the Model for End Stage Liver Disease score (MELD), complications like presence of fluid retention and hepatic encephalopathy; number of medication and diuretics; β-blockers and lactulose use were all compiled. The indications for liver transplantation were categorized into alcoholic cirrhosis, viral and other diseases.

In the second part of the study the patients evaluated in the pre-transplant who underwent transplantation were assessed in relation to the same parameters evaluated in the pre-transplant: nutritional, functional, metabolic, body composition, anthropometric, food intake and balance energy. For a description of the evolution of variables comparing the pre- and post-transplantation and evaluate the association of the variables evaluated the clinical outcomes of patients.

For the study about the prevalence of metabolic changes after liver transplantation in late post-transplant period, another population was evaluated. Patients undergoing liver transplantation between the years 2001-2014, which had data in medical records up to at least one year after surgery were included. To assess the prevalence and factors associated with hyperkalemia, information collected was: sex, age, underlying disease indication for transplantation, medication use, potassium, urea, creatinine and sodium values. Immunosuppressive drugs were: tacrolimus use and dose prescribed, and the residual dose; cyclosporine use and dose; prednisone use and dose. The use of other drugs included: furosemide, spironolactone, propranolol, captopril and enalapril.

To assess the prevalence of hypertension, diabetes and overweight according different doses of immunosuppression the presence of these conditions were collected from diagnosis described in the medical record of the patient, as well as the use of hypoglycemic agents and insulin medications will be evaluated; as well as the use of anti-hypertensive drugs. If the last weight registered in the medical record (post-transplant) subtracted from the weight recorded in the pre-transplant period will be considered. Those patients record that had water retention in the preoperative period, the estimated dry weight is considered. Those patients record that had water retention in the preoperative period, the estimated dry weight is considered. To do so, it will be contemplated from subtracting the estimated amount of liquid ascites and / or edema of the then current weight.

ELIGIBILITY:
Inclusion Criteria:

* Patients on the waiting list for liver transplant
* Over 20 years old
* Accepted the terms of survey

Exclusion Criteria:

* Under 20 years old
* Fulminant hepatitis
* Re-transplant
* Double transplant

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients on the waiting list for liver transplant at the University Hospital of University Federal of Minas Gerais.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2013-07 (Actual); Primary Completion 2017-10 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Nutritional status | December 2016
  Subjective Global Assessment

SECONDARY OUTCOMES:
Functional status | December 2016
  Dinamometry Heart rate variability Six minute walk test
Metabolic status | December 2016
  Resting Energy Expenditure Energetic Balance

OTHER OUTCOMES:
Metabolic status after liver transplantation | December 2016
  Hyperkalemia
Metabolic status long term after liver transplantation | December 2016
  Diabetes mellitus Hypertension Overweight

CONTACTS AND LOCATIONS:
Overall Officials: Helem Ribeiro, Principal Investigator — helemsena@gmail.com
Locations (1):
- Hospital of Clinics of the University Federal of Minas Gerais, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No